CLINICAL TRIAL: NCT02400853
Title: Research a New Predictive Marker of Intraventricular Hemorrhage in Very Preterm Infants: HEMO PREMA Study
Brief Title: Research a New Predictive Marker of Intraventricular Hemorrhage in Very Preterm Infants
Acronym: HEMO PREMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Purpose: Prevention
Other Study IDs: 2014/061/HP
Record Dates: First submitted 2015-03-02; First posted 2015-03-27 (Estimated); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Intraventricular Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- preterm infants with intracranial hemorrhage (Experimental): Cord blood analysis of preterm infants with radiological finding of intracranial hemorrhage, detected by ultrasound between day 5 and day 7 post-birth (Standard cranial echography) will be collected and analysed
  Interventions: Device: Standard cranial echography; Procedure: Cord blood analysis
- preterm infants without intracranial hemorrhage (Active Comparator): Cord blood analysis of preterm infants without radiological finding of intracranial hemorrhage, detected by ultrasound between day 5 and day 7 post-birth (Standard cranial echography) will be collected and analysed
  Interventions: Device: Standard cranial echography; Procedure: Cord blood analysis

INTERVENTIONS:
Device: Standard cranial echography — Standard cranial echography will be done at day 5 day 7 post-birth looking for radiological finding of intraventricular hemorrhage
Procedure: Cord blood analysis — Cord blood will be collected during deliverance and analysed

SUMMARY:
The most frequent complications in premature infants are neurological complications: intracranial hemorrhages and white matter lesions. In Epipage 2 study the incidence of severe intraventricular hemorrhages remains stable. Severe hemorrhages are associated with neurological sequelae.

A recent study in humans and in animals shows the role of the complex formed by plasminogen activator (t-PA) and its inhibitor (PAI-1) in the induction of vascular fragility via stromelysin (MMP-3). FIBRINAT study in Rouen University Hospital showed a rate of complex t-PA-PAI1 probably very high in preterm infants. An other factor maturation PDGF-C induced by t-PA is associated with the vascular embrittlement. Among the few genetic factors associated with cerebral palsy include 2 SNP of PAI-1 gene and one SNP in the gene of endothelial NO synthase.

The hypothesis is that a high rate of the complex t-PA-PAI-1 in cord blood could be a high risk of intracranial hemorrhage in preterm infants and provide predictive of their occurrence. The rates of MMP-3, PDGF-C and PAI-1 free in cord blood, and the polymorphism of PAI-1 gene and eNOS could separately or associated with the main criterion to identify predictive of hemorrhages.

The main objective is to search a rate difference of the complex t-PA-PAI-1 in cord blood of preterm infants (before 30 weeks of gestation) that would predict intracranial hemorrhage coming in the first days of life.

The secondary objectives are

* Evaluate potential marker risk of high levels of MMP-3, PAI-1 free, and PDGF-CC
* Search in both groups the presence of alleles -675G4 / G5 and 11053 (G / T) of the PAI-1 gene and -922 (A / G) of the eNOS gene.

  120 preterm infants will be included before 30 weeks of gestation with precise inclusion and exclusion criteria during a period of 3 years.

Patients will be divided into two groups according to whether they will or not showed intracranial hemorrhage (detected by ultrasound J5-J7).

The complex rate tPA-PAI-1, PAI-1 free, MMP-3 and PDGF-C will be measured. The comparison between the two groups will be carried out using statistical tests. Comparison of the presence of the alleles -675 4G and 11053T the PAI-1 gene or -922G eNOS gene between the two groups will be performed.

The demonstration of this hypothesis would permit to identify children from birth in whom the immediate implementation of preventive treatment of bleeding is desirable.

ELIGIBILITY:
Inclusion Criteria:

* Alive preterm infants between 24 weeks gestation and 29 weeks and 6 days
* Infants of both sexes
* Children whose parents signed a free and informed consent after oral information by one of the study investigators
* Exact term (pregnancy onset evaluated by the craniocaudal length or the date of the puncture in a medical assisted reproduction)
* Children with social protection

Exclusion Criteria:

* Maternal taking of antiplatelet therapy or anticoagulation within 48 hours of birth
* Acquired maternal disease constituting a risk factor for neonatal hemorrhage
* Constitutional maternal disease constituting a risk factor for neonatal hemorrhage
* Severe fetal malformation
* Cesarean birth after diagnosis of hydrocephalus detected in utero
* Minors parents
* History of mental disease,or sensory abnormality of one of the parents, which can lead to confusion about the study

Ages: 1 Day to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 175 (Actual)
Dates: Start 2015-07-10 (Actual); Primary Completion 2020-04-21 (Actual); Study Completion 2020-04-21 (Actual)

PRIMARY OUTCOMES:
tPA-PAI-1 Complex rate in cord blood | day 1
  tPA-PAI-1 Complex rate in cord blood will be analysed in the 2 groups of infants

SECONDARY OUTCOMES:
MMP-3 rate in cord blood | day 1
  MMP-3 rate in cord blood will be analysed in the 2 groups of infants
PAI-1 rate in cord blood | day 1
  PAI-1 rate in cord blood will be analysed in the 2 groups of infants
PDGF-CC rate in cord blood | day 1
  PDGF-CC rate in cord blood will be analysed in the 2 groups of infants
675G4 / G5 G11053T PAI-1 Genetic variations sequencing | day 1
  Polymorphism of specified sequence will be performed in the 2 groups of infants
A-922g eNOS Genetic variations sequencing | day 1
  Polymorphism of specified sequence will be performed in the 2 groups of infants

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane MARRET, Pr, Principal Investigator — UH Rouen
Locations (1):
- Rouen University Hospital, Rouen, France